CLINICAL TRIAL: NCT06027944
Title: More Than Meets the Eye? The Impact of Light on Mood Regulation in Humans
Brief Title: Impact of Light on Mood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-71791
Record Dates: First submitted 2023-08-23; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scene (Experimental): High fidelity scene of nature emitted from a monitor
  Interventions: Other: Light exposure
- Scrambled scene (Active Comparator): The same pixels that are used to create the scene in the alternate arm will be randomly scrambled on the monitor
  Interventions: Other: Light exposure

INTERVENTIONS:
Other: Light exposure — Participants will be exposed to 15 minutes of each arm. They will be exposed twice and a randomized order (1/2/1/2 or 2/1/2/1)

SUMMARY:
The investigators are examining whether the content of a visual scene impacts the antidepressant effects of light or if this impact is solely mediated by the intensity of the light.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60
* Mild depressive symptomatology

Exclusion Criteria:

* No depressive symptomatology
* Severe depressive symptomatology
* Active or unstable medical condition
* Diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in mood | 15 minutes
  Change in subjective mood as recored by the Positive and Negative Affect Schedule (PANAS). The PANAS ranges 10-50 on a positive mood scale (higher = more positive) and 10-50 on a negative mood scale (higher = more negative)

SECONDARY OUTCOMES:
Change in fast brain electrical activity | 15 minutes
  Change in the beta power spectrum (12.5-30 Hz) of the electroencephalogram (brain waves, measured in microvolts)
Change in systolic blood pressure (SBP) | 15 minutes
  Change in SBP (mm Hg) as measured by finger plethysmography
Change in heart rate variability (HRV) | 15 minutes
  Shift in the ratio of the power of low frequency to high frequency components in heart rate variability
Change in sympathetic activity | 15 minutes
  Sympathetic activity will be imputed through the galvanic skin response (GSR). Change in skin conductance (the electrical activity on the skin) will be measured in microsiemens

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of data collection, cleaning, and publication, all experimental data will be made available via Dryad
Supporting Information: Study Protocol, Analytic Code
Time Frame: within three months of publication, no time limit